CLINICAL TRIAL: NCT00006916
Title: A Phase II Trial Of Conventional Radiation Therapy Followed By Intratumoral Bleomycin Delivered Using A Refillable, Sustained Release Device (IND# 46,592) For The Treatment Of Supratentorial Glioblastoma
Brief Title: Radiation Therapy Followed by Bleomycin in Treating Adult Patients With Newly Diagnosed Supratentorial Glioblastoma Multiforme
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-BR-0013; CDR0000068343
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2015-11

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Bleomycin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation therapy followed by bleomycin via Ommaya reservoir (Experimental): 60.0 Gy/30 fractions x 2.0 Gy. Then within 2-6 weeks after completion of radiation therapy or at the time a patient experiences disease progression during or immediately after completion of radiation therapy, if clinically feasible, a modified Ommaya reservoir is implanted with the delivery catheter in the tumor or tumor cyst/cavity. Bleomycin, 15 units per week, is then given via the Ommaya reservoir without interruption for a maximum of two years as long as there is no toxicity above grade 3 or evidence of disease progression.
  Interventions: Biological: bleomycin; Device: Ommaya reservoir; Radiation: radiation therapy

INTERVENTIONS:
Biological: bleomycin
Device: Ommaya reservoir
Radiation: radiation therapy — 60.0 Gy/30 fractions x 2.0 Gy. For the first 46 Gy/23 fractions the treatment volume should include the volume of contrast-enhancing lesion and surrounding edema on pre-operative CT/MRI scan plus a 2 centimeter margin. If no edema is present, the margin should be 2.5 cm. After 46.0 Gy, the tumor volume should include the contrast-enhancing lesion (without edema) on the pre-surgery MRI/CT scan plus a 2.5 centimeter margin.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy followed by bleomycin in treating adult patients who have newly diagnosed supratentorial glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the median survival time of patients with newly diagnosed supratentorial glioblastoma multiforme treated with radiotherapy followed by sustained release intratumoral bleomycin.
* Determine the feasibility of this regimen in these patients.

OUTLINE: This is a multicenter study.

Within 4 weeks after surgical resection, patients receive radiotherapy daily 5 days a week for 6 weeks.

Within 2-6 weeks after completion of radiotherapy or at disease progression during radiotherapy, patients undergo surgical implantation of a modified Ommaya reservoir within the central area of the tumor. Patients then receive sustained release bleomycin intratumorally via the reservoir once a week for up to 2 years in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 72 patients will be accrued for this study within 5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial glioblastoma multiforme (with areas of necrosis) by surgical biopsy or excision within 4 weeks of study
* Tumor and/or any associated edema limited to one hemisphere and unifocal
* No gross invasion of a ventricular surface
* Tumor accessible
* No other astrocytoma
* No multifocal or recurrent malignant glioma
* No disease below the tentorium or beyond the cranial vault

PATIENT CHARACTERISTICS:

Age:

* Adult

Performance status:

* Zubrod 0-1

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Hemoglobin at least 10 g/dL (transfusion allowed)
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* Serum glutamic-oxaloacetic transaminase (SGOT) or Serum glutamic-pyruvic transaminase (SGPT) no greater than 2 times normal

Renal:

* Blood Urea Nitrogen (BUN) no greater than 25 mg/dL
* Creatinine no greater than 1.5 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No hypersensitive or idiosyncratic reaction to bleomycin
* No other prior malignancies within the past 2 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix or urinary bladder
* No other major medical illness or psychiatric impairment that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for glioblastoma multiforme
* No prior radiosensitizer for glioblastoma multiforme

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the head or neck resulting in overlapping radiotherapy fields

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2001-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy A. Patchell, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (13):
- United States (13):
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Cancer Treatment Center, Wooster, Ohio
  - St. John Health System, Tulsa, Oklahoma
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy Followed by Bleomycin Via Ommaya Reservoir
Started | 19
Completed | 14 (Subjects with survival data for the primary analysis are considered to have completed the study.)
Not Completed | 5
Not completed — Device not inserted | 4
Not completed — Complication of device insertion | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy Followed by Bleomycin Via Ommaya Reservoir
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 59 [24 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: This study stopped accrual early with 19 subjects accrued out of 72 planned therefore no analyses were performed.
Time Frame: From randomization to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 18 months.
Arm/Group | Radiation Therapy Followed by Bleomycin Via Ommaya Reservoir
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events are reported for all subjects starting radiation therapy and/or bleomycin. Subjects experiencing more than one of a given SAE (serious adverse event) are counted only once for that SAE. The same methodology was applied for non-SAE adverse events (AE).
Arm/Group | Radiation Therapy Followed by Bleomycin Via Ommaya Reservoir
Serious Adverse Events (participants affected / at risk) | 5/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy Followed by Bleomycin Via Ommaya Reservoir (N=19)
Infection (document (Blood and lymphatic system disorders) | 1
Endocrine-Other (Endocrine disorders) | 1
Coagulation disorde (Investigations) | 1
Leucopenia NOS (Investigations) | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1
Convulsions NOS (Nervous system disorders) | 3
Neurologic-Other (Nervous system disorders) | 1
Speech disorder NEC (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Oedema NOS (Vascular disorders) | 1
Thrombosis NOS (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy Followed by Bleomycin Via Ommaya Reservoir (N=19)
Haemoglobin decreased (Blood and lymphatic system disorders) | 3
Earache (Ear and labyrinth disorders) | 1
Hearing-Other (Ear and labyrinth disorders) | 3
Dry eye NEC (Eye disorders) | 1
Ocular-Other (Eye disorders) | 4
Vision blurred (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting NOS (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 11
Pain-Other (General disorders) | 1
Syndromes-Other (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 3
Ecchymosis (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increas (Investigations) | 1
Aspartate aminotransferase incre (Investigations) | 1
Blood alkaline phosphatase NOS i (Investigations) | 1
Leucopenia NOS (Investigations) | 1
Neutropenia (Investigations) | 1
Platelet count decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1
Amnesia NEC (Nervous system disorders) | 1
Convulsions NOS (Nervous system disorders) | 5
Depressed level of consciousness (Nervous system disorders) | 2
Dizziness (exc vertigo) (Nervous system disorders) | 1
Headache NOS (Nervous system disorders) | 5
Neurologic-Other (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Speech disorder NEC (Nervous system disorders) | 4
Taste disturbance (Nervous system disorders) | 3
Anxiety NEC (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Depression NEC (Psychiatric disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Skin-Other (Skin and subcutaneous tissue disorders) | 1
Oedema NOS (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
This study stopped accrual early due unmet targeted accrual goals with 19 subjects accrued out of 72 planned. No efficacy analyses were performed since the small number of patients would not have provided meaningful results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No